CLINICAL TRIAL: NCT01258478
Title: Short-Term Pre-operative Rehabilitation for Patients With Lung Cancer: A Randomized Trial.
Brief Title: Lung Cancer Rehabilitation Study
Acronym: LCRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Dr. Pierre-Olivier Bridevaux, University Hospital Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocole 09-263
Record Dates: First submitted 2010-12-07; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC, rehabilitation, CPET, lung resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rehabilitation (Experimental): Three weeks of outpatient, intensive physical rehabilitation before lung resection surgery.
  Interventions: Other: Rehabilitation
- usual care (Sham Comparator): Usual care before surgery is provided
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Rehabilitation — Three weeks of outpatient, intensive physical rehabilitation before lung resection surgery.
  Arms: rehabilitation
Other: Usual care — Usual care
  Arms: usual care

SUMMARY:
Patients suffering from non small cell lung cancer(NSCLC), depend upon lung removal to increase their chances of survival. But, this type of surgery cannot be advised to patients with significant heart disease, limited lung fuction or reduced physical fitness. Intensive physical training has been shown to increase aerobic fitness in healthy subjects.

The purpose of this study is to determine the effect of a short term rehabilitation prior to surgery on the post-operative and physiological outcomes for patients undergoing this type of surgery.

DETAILED DESCRIPTION:
For patients with non small cell lung cancer (NSCLC), lung resection surgery is the only treatment option which increases survival. However, surgery can not be offered to those with significant heart disease, limited lung function or lacking physical fitness. These are all major risk factors for operative outcome. Cardio-pulmonary exercise testing (CPET) allows direct measurement of aerobic physical fitness through maximal oxygen consumption (VO2 max). A recent update of professional guidelines (ERS/ESTS) has emphasized the importance of CPET in preoperative risk stratification of patients with NSCLC. Interestingly, intensive physical training has been shown to increase aerobic fitness in animals and healthy subjects whereas improvement of VO2 max has been observed in preliminary pilot studies conducted in patients undergoing surgery for NSCLC. However, the net effect of short-term, intensive, outpatient rehabilitation on clinically relevant outcomes, such as major post-operative cardio-pulmonary complications, as well as physiological outcomes is unknown.

Objectives:

1. To assess the physiological effect of 3 weeks of intensive physical training in patients eligible for NSCLC surgery.
2. To assess the effect of physical training on post-operative outcomes.
3. To identify the clinical variables, laboratory tests and specific gene polymorphisms (SNPs) associated with these outcomes.

ELIGIBILITY:
Inclusion Criteria:

Proven or suspected lung cancer, stage III A or less (eligible for surgical cure), documented by CT-scan or Positron Emission Tomography CT scan (PET-CT)

Exclusion Criteria:

* Contra-indication to perform cardio-pulmonary exercise test (uncontrolled cardiac disease, severe pulmonary hypertension, osteo-articular limitations impeding cycling)
* Inability to adhere to rehabilitation program (because of clinically limiting comorbidity, psychiatric condition or osteoarthritis)
* Clinically limiting or untreated heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
A composite endpoint of respiratory or cardiac or other post-operative complications requiring therapy | 30 days after surgery
  Respiratory Pneumonia Atelectasis (requiring bronchoscopy or positive expiratory pressure) Mechanical ventilation >12 hours Unplanned re-intubation Acute lung injury or acute respiratory distress syndrome (ALI/ARDS) Cardiac Acute heart failure Myocardial infarction or acute coronary syndrome Arrhythmia Other Delirium, mental status changes Stroke or transient ischemic accident 30-day mortality Acute renal failure (doubling of baseline pre-operative value) Surgical site infection

SECONDARY OUTCOMES:
All endpoints in primary outcomes, taken separately and others, mentioned below | 1 year
  90 day mortality Hospital Length of stay, admission and re-admission in ICU Surgical wound infections Quality of life scores CPET and other physiological tests changes from baseline to week 3 Echocardiography changes from baseline to week 3, limited to those with high baseline NT-pro-BNP value (>300 ug/L) or those with a Lee score ≥2 Non invasive measurement of tissue oxygenation using Near Infrared Spectroscopy (NIRS) Nutritional status changes from baseline to week 3 Smoking behaviour changes from baseline to week 3 Cardiac autonomic nervous control

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Karenovics W, Licker M, Ellenberger C, Christodoulou M, Diaper J, Bhatia C, Robert J, Bridevaux PO, Triponez F. Short-term preoperative exercise therapy does not improve long-term outcome after lung cancer surgery: a randomized controlled study. Eur J Cardiothorac Surg. 2017 Jul 1;52(1):47-54. doi: 10.1093/ejcts/ezx030. PMID 28419206
- [Derived] Licker M, Karenovics W, Diaper J, Fresard I, Triponez F, Ellenberger C, Schorer R, Kayser B, Bridevaux PO. Short-Term Preoperative High-Intensity Interval Training in Patients Awaiting Lung Cancer Surgery: A Randomized Controlled Trial. J Thorac Oncol. 2017 Feb;12(2):323-333. doi: 10.1016/j.jtho.2016.09.125. Epub 2016 Oct 19. PMID 27771425